CLINICAL TRIAL: NCT03890094
Title: Safety and Efficacy of Sufentanil Combined With Midazolam in Bronchoscopy Under Conscious Sedation: Retrospective Study
Status: Completed | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, ShiYue Li, Clinical Professor, Guangzhou Institute of Respiratory Disease
Other Study IDs: Suretro2013
Record Dates: First submitted 2019-03-24; First posted 2019-03-26 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Bronchoscopy; Sedation
Keywords: Sufentanil; Bronchoscopy; Conscious sedation; midazolam
MeSH Terms: interventions — Sufentanil

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Sufentanil and Midazolam: Patients who had undergone bronchoscopy applying topical lidocaine, sufentanil and midazolam under conscious sedation in the First Affiliated Hospital of Guangzhou Medical University from September 2013 to July 2017 were included in this study.
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Sufentanil — Patients were applied sufentanil and midazolam intravenously and topical anesthetized.

SUMMARY:
The aim of this study was to determine the safety and efficacy of sufentanil combined with midazolam in bronchoscopy under conscious sedation. A retrospective analysis was conducted on all patients undergoing bronchoscopy applying sufentanil and midazolam under conscious sedation in the First Affiliated Hospital of Guangzhou Medical University from September 2013 to July 2017.

ELIGIBILITY:
Inclusion Criteria:

Patients who had undergone bronchoscopy applying topical lidocaine, sufentanil and midazolam under conscious sedation in the First Affiliated Hospital of Guangzhou Medical University from September 2013 to July 2017

Exclusion Criteria:

Patients who had undergone bronchoscopy not applying topical lidocaine, sufentanil and midazolam under conscious sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: According to guidelines of bronchoscopy, patients had no food by mouth for 4h and to allow clear fluids by mouth up to 2 h before bronchoscopy. Oxygen supplementation was given to the patients through the nasal cannula (2-5L/min, adjusted as needed). 2% lidocaine was applied for topical anesthesia. Sufentanil and midazolam were applied intravenously.
Sampling Method: Probability Sample
Enrollment: 11158 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Oxygen desaturation | during the procedure
  Percentage of patients whose oxygen saturation decreased to lower than 80% during procedure

CONTACTS AND LOCATIONS:
Overall Officials: Shiyue Li, Professor, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No